CLINICAL TRIAL: NCT00220480
Title: A Naturalistic Study of the Efficacy and Safety of Escitalopram in Treatment Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Chaim Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-04-3434-JZ-CTIL
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: escitalopram — 10 to 30 mg / day

SUMMARY:
The primary objective of this multicenter study is to evaluate the efficacy of escitalopram in treatment resistant depression (TRD), assessed by 2 consecutive failed antidepressant treatments from different classes. The last treatment received is a 6 week prospective trial with venlafaxine.

ELIGIBILITY:
Inclusion Criteria:

Any patient who meets all of the following criteria is eligible for inclusion in the Prospective phase I of the study:

1. The patient is able to read and understand the patient information sheet.
2. Prior to any screening procedures, the patient must have signed the informed consent form. No study-related procedures may be performed before the patient has signed the form.
3. The patient is an in- or outpatient, male or female.
4. The patient is between 18 and 65 years of age.
5. The patient suffers from a diagnosis of recurrent Major Depressive Disorder (current episode assessed with the MINI), moderate or severe, according to DSM-IV-TR criteria (classification code = 296.3x).
6. The patient has a total score of 22 or higher on the MADRS.
7. The patient has been treated for the current episode with an antidepressant (other than escitalopram or venlafaxine) prescribed continuously at the optimal dose (see table Appendix 1) for at least the 4 weeks preceding selection (AD1).
8. The investigator considers switching treatment to venlafaxine (AD2), prescribing it at its optimal dose, defined by the study protocol.

Exclusion Criteria:

Any patient who meets one or more of the following criteria cannot be included in the screening phase of the study:

1. The patient has previously participated in this study.
2. Results from blood sampling at selection show for the antidepressant prescribed (AD1), that plasma concentration is below the expected threshold according to time of last intake.
3. The patient has taken another antidepressant in combination to the antidepressant to which he/she is considered as non-responder (AD1).
4. The patient has one or more of the following conditions:

   1. Any current psychiatric disorder established as the principal diagnosis other than Major depressive episode as defined in the DSM-IV-TR (assessed with the MINI).
   2. Any Substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR.
   3. Any severe personality disorder according to investigator clinical judgement, that might compromise the study.
5. The patient uses disallowed recent or concomitant medication within the specified time periods:

   1. oral antipsychotic drugs within 2 months and depot antipsychotic preparations within the past 6 months.
   2. ECT within the past 6 months.
   3. lithium, carbamazepine, valproate or valpromide within the past month.
   4. any benzodiazepines at a dose higher than 10 mg diazepam or equivalent, within the last week.
   5. any non-benzodiazepine anxiolytics within the last week.
   6. serotonin agonists within the last week.
   7. any other drug with potential psychotropic effects within the last week.
   8. any drug known to lower blood pressure in the last week.
6. The patient has been treated with any investigational product within 3 months prior to screening.
7. The patient has been treated during the current episode with escitalopram or venlafaxine.
8. The patient has a history of severe drug allergy or hypersensitivity, or known hypersensitivity to escitalopram or venlafaxine.
9. The patient started (or will start) formal psychotherapy in the month preceding inclusion.
10. The patient has a previous history of convulsive disorder other than a single childhood febrile seizure.
11. The patient presents evidence of urinary retention or glaucoma.
12. The patient has a serious illness and/or serious sequelae thereof, including liver or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic, or metabolic disturbance.
13. The patient has, in the opinion of the investigator, on the basis of a physical examination, medical history and vital signs, a comorbid conditions(s) that would render inclusion in the study unsafe.
14. The patient takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy.
15. The patient, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-02; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
MADRS | 8 to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University
Locations (4):
- Israel (4):
  - Rambam Medical Center, Haifa
  - Ness Ziona Mental Health Center, Ness Ziona
  - Gehah Mental Health Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan